CLINICAL TRIAL: NCT06723041
Title: Acupressure for Anxiety: A Randomized Controlled Trial of an Acupressure Intervention for Patients Receiving Cancer-Directed Therapy
Brief Title: Acupressure for the Reduction of Anxiety in Patients Receiving Cancer-Directed Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-007105; NCI-2024-09813 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-007105 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Acupressure; Health Promotion; Educational Status

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are blinded during intervention only and unblinded following intervention completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (true acupressure) (Experimental): Patients undergo true acupressure over 10 minutes on study. Patients that choose to learn self-administration acupressure at home receive educational information and undergo self-administration acupressure sessions at least BID for seven days.
  Interventions: Procedure: Acupressure Therapy; Procedure: Acupressure Therapy - self-administered; Other: Health Promotion and Education; Other: Survey Administration
- Arm II (sham acupressure) (Sham Comparator): Patients undergo sham acupressure over 10 minutes on study. Patients that choose to learn self-administration acupressure at home receive educational information and undergo self-administration acupressure sessions at least BID for seven days.
  Interventions: Procedure: Acupressure Therapy - placebo; Procedure: Acupressure Therapy - self-administered; Other: Health Promotion and Education; Other: Survey Administration

INTERVENTIONS:
Procedure: Acupressure Therapy — Undergo true acupressure
  Other Names: Acupressure; Ischemic Compression
  Arms: Arm I (true acupressure)
Procedure: Acupressure Therapy - placebo — Undergo sham acupressure
  Other Names: Acupressure; Ischemic Compression
  Arms: Arm II (sham acupressure)
Procedure: Acupressure Therapy - self-administered — Undergo self-administered acupressure
  Other Names: Acupressure; Ischemic Compression
Other: Health Promotion and Education — Receive educational handouts
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinicaI trial is being done to determine if acupressure is helpful to reduce anxiety related to chemotherapy, compared with "sham" (or placebo) acupressure in patients with cancer. Anxiety, experienced by many patients with cancer, can be related to chemotherapy and may contribute to other symptoms, such as nausea and poor quality of life. Some patients diagnosed with cancer express interest in non-medicine ways to manage symptoms. Acupressure is the application of non-invasive finger pressure along energy points throughout the body in order to relieve pain and induce a feeling of well-being. Previous research has shown that acupressure can help both adults and children with their anxiety in certain situations, such as after surgery. Patients can be taught how to do the acupressure on themselves, making this an intervention that can be done anywhere. Acupressure is well tolerated with minimal reports of adverse reactions. Undergoing acupressure may be effective in reducing anxiety in cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To test the efficacy of a nurse-applied acupressure intervention for anxiety associated with active cancer-directed therapy.

SECONDARY OBJECTIVES:

I. To test the efficacy of a patient-applied acupressure intervention for anxiety associated with active cancer-directed therapy.

II. To assess whether acupressure appears to improve nausea related to cancer and cancer-directed therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo true acupressure over 10 minutes on study. Patients that choose to learn self-administration acupressure at home receive educational information and undergo self-administration acupressure sessions at least twice daily (BID) for seven days.

ARM II: Patients undergo sham acupressure over 10 minutes on study. Patients that choose to learn self-administration acupressure at home receive educational information and undergo self-administration acupressure sessions at least BID for seven days.

ELIGIBILITY:
Inclusion Criteria:

* NURSE-LED INTERVENTION: Age >= 18 years and be diagnosed with cancer
* NURSE-LED INTERVENTION: Undergoing systemic, antineoplastic therapy
* NURSE-LED INTERVENTION: Ability to provide oral consent
* NURSE-LED INTERVENTION: Willingness to undergo a nurse-led acupressure intervention
* NURSE-LED INTERVENTION: Willingness and ability to complete pre- and post-intervention questionnaires in English
* NURSE-LED INTERVENTION: Report acute anxiety as a 5 or higher on a scale for 0 (no anxiety) to 10 (severe anxiety)
* SELF-ADMINISTRATION INTERVENTION: Age >= 18 years and be diagnosed with cancer
* SELF-ADMINISTRATION INTERVENTION: Undergoing systemic, antineoplastic therapy
* SELF-ADMINISTRATION INTERVENTION: Ability to provide oral consent
* SELF-ADMINISTRATION INTERVENTION: Willingness to undergo a nurse-led acupressure intervention
* SELF-ADMINISTRATION INTERVENTION: Willingness and ability to complete pre- and post-intervention questionnaires in English
* SELF-ADMINISTRATION INTERVENTION: Report acute anxiety as a 5 or higher on a scale for 0 (no anxiety) to 10 (severe anxiety)
* SELF-ADMINISTRATION INTERVENTION: Reports 2+/day anxiety episodes at home
* SELF-ADMINISTRATION INTERVENTION: Interested in learning self-administered acupressure

Exclusion Criteria:

* Prior experiences with acupressure, or training in acupressure points

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in acute anxiety | Up to 2 weeks
  Will be compared between treatment groups. This will be measured by changes in responses to a single item, "Please rate the following symptoms, based on how you feel at the current time (please indicate the one most correct response)," with responses provided on a Likert scale from 0 (no anxiety) to 10 (worst possible anxiety).

SECONDARY OUTCOMES:
Associations between changes in anxiety and demographic variables | Up to 2 weeks
  Demographic variables, including age, gender identity, race/ethnicity, cancer type, cancer stage, and cancer therapy type, will be compared with answers to anxiety question specified in Outcome 1.
Efficacy of self-administered acupressure | Up to 2 weeks
  Assessed by the number of participants in each arm (true vs sham) who are willing to complete self-administered acupressure.
Changes in anxiety-related symptoms | Up to 2 weeks
  Assessed using an anxiety questionnaire administered at baseline and post-intervention. Seven items (anxiety, nausea, pain, wellbeing, relaxation, worry, and distress) are rated on a scale of 0 (strongly disagree) to 10 (strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Cathcart-Rake, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials